CLINICAL TRIAL: NCT02567279
Title: Impact of Denosumab in the Prevention of Bone Loss in Non-menopausal Women With Anorexia Nervosa
Acronym: DIBLAN
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Great difficulties were encountered during recruitment, for fear Denozumab. Only 2 patients have been included since the study start.
Sponsor: University Hospital, Montpellier (Other)
Collaborators: University Hospital, Lille (Other); Nantes University Hospital (Other); University Hospital, Paris (Other); University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 9531
Record Dates: First submitted 2015-10-01; First posted 2015-10-02 (Estimated); Last update posted 2019-01-07 (Actual); Status verified 2019-01

CONDITIONS: Anorexia Nervosa
MeSH Terms: conditions — Anorexia Nervosa | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Denosumab subcutaneous injections (Active Comparator): The treated group (n = 42) will receive Denosumab (60 mg, two subcutaneous injections at M0 and M6) associated with a daily treatment of vitamin D (800 IU) + calcium (1000 mg).
  Interventions: Drug: Denosumab subcutaneous injections
- Placebo subcutaneous injections (Placebo Comparator): The control group (n = 42) will received a placebo injection (two subcutaneous injections at M0 and M6) with daily treatment of vitamin D (800 IU) +calcium (1000 mg).
  Interventions: Drug: Placebo subcutaneous injections

INTERVENTIONS:
Drug: Denosumab subcutaneous injections — Subcutaneous injection of Denosumab 60 mg, one injection at baseline and another injection at 6 months
  Other Names: Treated group
  Arms: Denosumab subcutaneous injections
Drug: Placebo subcutaneous injections — Subcutaneous injection of Placebo, one injection at baseline and another injection at 6 months
  Other Names: Control group
  Arms: Placebo subcutaneous injections

SUMMARY:
The drastic reduction of nutritional intake in anorexia nervosa(AN) alters many hormonal factors that regulate the activity of bone cells. This alteration of bone remodeling is characterized by increased bone resorption and decreased bone formation, leading to a marked reduction of bone mineral density, osteoporosis and an increased risk of fracture.

To date, there is a paucity of studies and no consensus on the management of bone loss in patients with AN. The few previous studies were performed with small samples and using short follow-up periods.

Denosumab is a fully human monoclonal antibody that binds with high specificity to human RANKL (6, 7), thereby reducing the number and activity of osteoclasts and therefore decreasing bone resorption that was found increased in patients AN.

Denosumab may transiently protect bone whilst psychonutritional management will induce a weight restoration

DETAILED DESCRIPTION:
The project propose to assess, with a double-blind multicentric randomized clinical trial, the effects of Denosumab on bone mineral density (BMD) change at lumbar spine over 12 months among patients suffering from an acute anorexia nervosa (AN).

84 patients suffering from a current anorexia nervosa with an evidence of low BMD determined by a Z-score value < -2 DS at least one site (lumbar spine or total proximal femur) will be recruit .

Eligible patients will be randomized into two groups: denosumab versus placebo. Each patient will attend a total of 8 scheduled visits, which will be completed over a period of 24 months +/- 15days from screening visit to end of study (inclusion, 10 days, and 3, 6, 12, 15, 18, & 24 months).

ELIGIBILITY:
Inclusion criteria:

* Patients with a current AN defined by DSM-V criteria
* Being female
* Age over or equal to 18 years and less or equal to 40 years

  . For patients under 20 years of age, effective bone maturation (attested by a radiography of the hip)
* Agree to take contraception up to five months after the last injection of denosumab .
* Absence of pregnancy evidenced by an interview and a negative assay of human chorionic gonadotropin (ßhCG).
* Evidence of low BMD determined by Z-score value < -2 DS (at least one site (lumbar spine or total proximal femur)
* Signing an informed consent.

Exclusion criteria:

* Not affiliated to a social security scheme or not being the beneficiary of such a scheme.
* Severe hepatic cytolysis with transaminase up to 5 times normal.
* Severe dental problems: in case of doubt an assessment by a dentist will be required before inclusion.
* Desire of pregnancy during the two years of follow-up study.
* Disease or treatment potentially responsible for secondary osteoporosis.
* Participant already treated with a molecule known to have an effect on bone
* Diabetes.
* Current hypocalcemia.
* Immunodeficiency.
* Cancer with bone lesions
* Patient on protectice measures (guardianship or trusteeship)
* Hypersensitivity to the active substance or to any of the excipients of Prolia®
* Unable to read and / or write and understand the methodology of the study
* Reporting relationship to the investigator
* Anticipate a long stay outside the region that would prevent compliance with the schedule of visits
* Participation to other biomedical research on health products
* Deprived of liberty
* Breastfeeding

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2019-01-03 (Actual); Study Completion 2019-01-03 (Actual)

PRIMARY OUTCOMES:
Value of bone mineral density in lumbar spine (g/cm2) | 12 months
  Comparison of bone mineral density changes in the lumbar spine at M12 between groups with Denosumab and placebo after two injections either of Denosumab or placebo. Bone mineral density is objectified by the Z-score obtained by bone mineral density.

SECONDARY OUTCOMES:
value of bone mineral density in the whole body, the total proximal femur and the radius (g/cm2) | 12 months
  Comparison of bone mineral density changes in the whole body, the total proximal femur and the radius between groups at M12 after two injections of Denosumab.
values of bone mineral density at 24 months | 24 months
  Comparison of the levels of bone mineral density at 24 months
values of bone remodeling markers at 24 months | 24 months
  Comparison of the values of bone remodeling markers at 24 months
links between ESR1 genotype and bone minéral density at Baseline and response to Denosunab | 12 months
  Assess the links between ESR1 genotype and BMD at baseline and response to Denosunab (variation of BMD between baseline and 12 months).

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien Guillaume, MD PhD, Principal Investigator — Hôpital Lapeyronie - CHU de Montpellier
Locations (1):
- CHU Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No